CLINICAL TRIAL: NCT06729996
Title: Randomized, Parallel Group, Dose Escalation Trial of Pioglitazone Versus Empagliflozin for Chronic Pancreatitis/Recurrent Acute Pancreatitis Associated Diabetes Mellitus: The PEP-DM Trial
Brief Title: Pioglitazone Versus Empagliflozin for Chronic Pancreatitis/Recurrent Acute Pancreatitis Associated Diabetes Mellitus
Acronym: PEP-DM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Yogish C. Kudva, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-003868
Record Dates: First submitted 2024-12-05; First posted 2024-12-12 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pancreatitis, Chronic; Pancreatitis, Acute; Diabetes Mellitus
Keywords: pancreatitis; diabetes; diabetes mellitus; empagliflozin; pioglitazone
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Diabetes Mellitus | interventions — Pioglitazone; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (PIO) (Experimental): PIO (Actos) is a thiazolidinedione and an agonist for peroxisome proliferator activated receptor (PPAR) gamma indicated as an adjunct to diet and exercise to improve glycemic control in adults with type 2 DM in multiple clinical settings. Its use has limitation for type 1 DM or for treatment of diabetic ketoacidosis. It is contraindicated to use in established NYHA class III or IV heart failure.
  Interventions: Drug: Pioglitazone (PIO)
- Empagliflozin (EMPA) (Experimental): EMPA is a sodium-glucose co-transporter 2 inhibitor, FDA approved drug. It is indicated to reduce the risk of cardiovascular death and hospitalization for heart failure in adults with heart failure, to reduce the risk of cardiovascular death in adults with type 2 DM and established cardiovascular disease and as an adjunct to diet and exercise to improve glycemic control in adults with type 2 DM. It is not recommended in patients with type 1 DM. It may increase the risk of diabetic ketoacidosis. Not recommended for use to improve glycemic control in adults with type 2 DM with an eGFR less than 30mL/min/1.73m2.
  Interventions: Drug: Empagliflozin (EMPA)

INTERVENTIONS:
Drug: Pioglitazone (PIO) — Subjects will take 30 mg tablet, once daily in the morning, taken with or without food for 12 weeks and after 12 weeks dose will be escalated to 45 mg based on Hemoglobin A1c (HbA1c) levels (HbA1c >7.0% at 12 weeks, escalate the dose) once daily in the morning, taken with or without food till 24 weeks.
  Arms: Pioglitazone (PIO)
Drug: Empagliflozin (EMPA) — Subjects will start with 10 mg dose, once daily in the morning, taken with or without food for 12 weeks and after 12 weeks dose will be escalated to 25 mg based on Hemoglobin A1c (HbA1c) levels (HbA1c >7.0% at 12 weeks, escalate the dose) once daily in the morning, taken with or without food.
  Arms: Empagliflozin (EMPA)

SUMMARY:
The purpose of this study is to evaluate efficacy of pioglitazone (PIO) versus empagliflozin (EMPA) to improve glycemic control in people with Chronic Pancreatitis (CP) or Recurrent Acute Pancreatitis (RAP) associated with Diabetes Mellitus (DM). To evaluate mixed meal response in PIO versus EMPA group to better understand physiology of both therapies in CP-DM.

DETAILED DESCRIPTION:
This trial will test the efficacy of PIO versus EMPA in improving glycemic control in CP-DM. The anticipated enrollment will consist of 40 subjects, age 18-70 years who have been diagnosed with CP or RAP with DM, at two clinical sites in the United States. The primary objective is to evaluate the efficacy of PIO vs. EMPA to improve glycemic control in people with CP or RAP associated with DM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18-70 years at the time of enrollment.
* RAP or CP with DM diagnosed before or after CP diagnosis (Confirmed CP on imaging or RAP based on PROCEED study criteria, and confirmed DM as per ADA criteria or clinically diagnosed with DM and on antihyperglycemic therapy)
* Able to provide written informed consent and participate in longitudinal follow-up
* Stable last annual retinal exam within 1 year prior to enrollment.
* HbA1c level 7-10% at screening visit.
* Fasting plasma glucose <220 mg/dL at screening visit.
* Not on any antihyperglycemic medication except Metformin
* Willing to perform blood glucose and ketone testing on study provided meters as per study protocol.

Exclusion Criteria:

* Inability to take PIO or EMPA due to prior hypersensitivity or allergic reaction or current use of medications with potential for drug-drug interactions (Pioglitazone: Drug information - UpToDate, Empagliflozin: Drug information - UpToDate)
* Diagnosed with Type 1 Diabetes
* Pregnancy or lactation in women (positive urine pregnancy test at screening will lead to exclusion)
* History of bleeding disorders (e.g., Hemophilia A (factor VIII deficiency), hemophilia B (factor IX deficiency), von Willebrand disease, platelet disorders etc)
* Presence of hepatic impairment, ALT >3 x ULN with no etiology known at the time of enrollment or any evidence of acute/chronic liver disease
* Ongoing treatment for any malignancy requiring systemic treatment (non-melanoma skin cancers treated in dermatologists' office would be acceptable)
* Presence of osteoporosis (the threshold of bone density value below the -2.5 SDS of T-score or presence of one or more fragility fractures), on electronic medical record.
* Recent inflammatory illness within the 30 days preceding enrollment (e.g.: URTI, episode of AP, etc)
* History of heart failure classified by New York Heart Association as Class III or greater
* History of kidney dysfunction classified by eGFR of <30 mL/min/min
* Participation in any clinical trial within 30 days before screening for an approved or non-approved investigational medical product.
* Active alcohol dependence or chemical dependence including tobacco based on investigator discretion
* On a ketogenic diet
* Autoimmune pancreatitis, obstructive pancreatitis, and prior surgery of pancreas
* Any condition which could jeopardize participant safety as per investigator opinion, (hemolytic anemia limiting HbA1c reliability, any evidence of fluid overload, presence of Congestive heart failure etc).
* Recent DKA or signs of decompensated diabetes in last 6 months or increased β hydroxybutyrate levels (>0.4 mmol/L) at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | Baseline to 24 weeks
  Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An HbA1C level below 5.7 percent is considered normal. Reported as percentage of glycated hemoglobin
Area under curve (AUC) for glucose | Baseline to 24 weeks
  Pre-post study difference in AUC for glucose
AUC for C-peptide | Baseline to 24 weeks
  Pre-post study difference in AUC for C-Peptide
AUC for Insulin | Baseline to 24 weeks
  Pre-post study difference in AUC for Insulin
AUC for glucagon | Baseline to 24 weeks
  Pre-post study difference in AUC for glucagon

SECONDARY OUTCOMES:
Fasting plasma glucose | Baseline to 24 weeks
  Pre-post study difference in Fasting plasma glucose
Lean mass | Baseline to 24 weeks
  Pre-post study difference in lean mass
Fat mass | Baseline to 24 weeks
  Pre-post study difference in fat mass
Visceral fat | Baseline to 24 weeks
  Pre-post study difference in visceral fat
Fecal elastase | Baseline to 24 weeks
  Pre-post study difference in Fecal elastase (ELISA quantitative test, normal >200 mcg/g)
High Sensitivity C-Reactive Protein (Hs-CRP) | Baseline to 24 weeks
  Pre-post study difference in Hs-CRP
Total cholesterol, LDL, HDL and Triglyceride | Baseline to 24 weeks
  Pre-post study difference in Total cholesterol, LDL, HDL and Triglyceride
β-Hydroxybutyrate | Baseline to 24 weeks
  Pre-post study difference in β-Hydroxybutyrate
Body weight | Baseline to 24 weeks
  Pre-post study difference in body weight
Blood Pressure | Baseline to 24 weeks
  Pre-post study difference in Blood Pressure
Body Mass Index (BMI) | Baseline to 24 weeks
  Pre-post study difference in BMI
Patient-Reported Outcomes Measurement Information System - 29 Profile v2.1 (PROMIS-29 Profile v2.1) | Baseline to 24 weeks
  The PROMIS-29 Profile assesses following domains:
  * Physical function
  * Pain interference
  * Anxiety
  * Depression
  * Fatigue
  * Sleep disturbance
  * Ability to participate in social roles and activities
  PROMIS-29 is scored using T-scores. Higher T-scores indicate a higher level of the underlying construct.
  Each domain has a set of questions, typically 4 to 6 items, and responses are rated on a 5-point Likert scale (e.g., "Never," "Rarely," "Sometimes," "Often," "Always" or "Not at all," "A little bit," "Somewhat," etc.). The responses are then scored on a T-score scale (with a mean of 50 and a standard deviation of 10 in the general population).
  T-scores Interpretation:
  * A T-score of 50 is the average score for the general population.
  * T-scores above 50 indicate better functioning or less severe symptoms.
  * T-scores below 50 indicate worse functioning or more severe symptoms.
Insulin sensitivity | Baseline to 24 weeks
  Change in sensitivity from baseline vs 24 weeks (Homeostatic Model Assessment, Matsuda Index)
Beta cell function | Baseline to 24 weeks
  Change in Beta cell function from baseline vs 24 weeks using oral disposition index

OTHER OUTCOMES:
Ketosis | Baseline to 24 weeks
  Percentage of participants experiencing Ketosis based on meter data
Diabetic Ketoacidosis (DKA) events | Baseline to 24 weeks
  Number of DKA events
Insulin needs | Baseline to 24 weeks
  Percentage of participants experiencing requirement for insulin
Chronic pancreatitis exacerbation | Baseline to 24 weeks
  Percentage of participants experiencing CP exacerbation
Acute pancreatitis episodes | Baseline to 24 weeks
  Percentage of participants experiencing AP episodes
Exocrine pancreatic insufficiency | Baseline to 24 weeks
  Percentage of participants experiencing incident exocrine pancreatic insufficiency
Vitamin D | Baseline to 24 weeks
  Decrease in vitamin D
Bone fractures | Baseline to 24 weeks
  Percentage of participants experiencing bone fractures
Adverse events | Baseline to 24 weeks
  Adverse events: Anemia, edema, urinary tract infection, Vaginal yeast infection

CONTACTS AND LOCATIONS:
Overall Officials: Yogish Kudva, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No